CLINICAL TRIAL: NCT05965817
Title: Fluorescence-guided Resection Of Colorectal Liver Metastases Using SGM-101 and Indocyanine GREEN
Acronym: FOCUS GREEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, MD, PhD, principle investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P23
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer; Liver Metastasis Colon Cancer; Image
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: In total 10 patients will be included who are scheduled for resection of colorectal liver metastases and meet at least one of the following criteria:
  1. Scheduled for resection of >3 CRLM or,
  2. Completed neo-adjuvant chemotherapy, of which the last course was completed within 3 months before surgery or,
  3. Scheduled for surgery because of a locally recurrent liver metastasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with colorectal liver metastases receiving SGM-101 and ICG (Experimental): In total 10 patients will be included who are scheduled for resection of colorectal liver metastases and receive SGM-101 and ICG
  Interventions: Drug: SGM-101 op top of ICG

INTERVENTIONS:
Drug: SGM-101 op top of ICG — SGM-101 op top of ICG

SUMMARY:
This will be the first trial testing the feasibility of working simultaneously with the two fluorescent dyes ICG and SGM-101 in 10 patients with colorectal metastases.

DETAILED DESCRIPTION:
25-30% of patients with colorectal cancer develop colorectal liver metastases (CRLM). Cornerstone for optimal survival is achieving radical surgical resections of all metastases . To assist the surgeon in achieving this, the use of intra-operative ICG for fluorescent tumour delineation has widely been adopted as standard of care. Multiple international trials have demonstrated that the use of ICG increases the rate of radical resections and result in the detection of additional malignant lesions invisible to the naked eye. However, the rate of false positives is still high and although it has increased the number of radical resections, even in a minimal invasive cohort the unintended R1 rate is still as much as 8%. Therefore, there is a need of an additional real-time intra-operative tool to detect R1 resections, especially in patients with a priori high risk for R1. To illustrate, in a large shared database of the Erasmus University Medical Center was found that patients that either received neoadjuvant chemotherapy, underwent a resection for >3 CRLM or patients that had a locally recurrent liver metastasis were independently associated with high R1 rates, ranging between 23-29%. Therefore, here is proposed the addition of SGM-101, a tumour targeted (carcinoembryonic antigen, CEA) NIR-fluorescence probe to ICG in patients scheduled for a resection with high risk of R1, ultimately to reduce the R1 ratio. This is the first trial testing the feasibility of working simultaneously with the two fluorescent dyes. If feasibility is met in this trial, this is a step-up towards a powered trial with primary objective to reduce the rate of R1 resections.

An additional exploratory objective of this study is to investigate the feasibility of SGM-101's potential to isolate circulating tumour cells (CTCs) and tumour-derived extracellular vesicles (EVs) as biomarkers for CRC. The load of CTCs and EVs in the circulation is strongly associated with poor clinical outcomes. Studies have shown that they contain information about the molecular profile of the tumour. The administration of SGM-101 may enable the detection of CEA positive CTCs and EVs.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  1. Diagnosed with liver metastases of colorectal origin for which surgical resection is proposed and meet at least one of the following criteria:

     1. Scheduled for surgical resection of >3 CRLM or;
     2. completed neo-adjuvant therapy, of which the last course was completed within 3 months before surgery or;
     3. Scheduled for surgery because of a locally recurrent liver metastasis.
  2. ≥18 years old.
  3. Willing and capable to give informed consent before study specific procedures

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:

  1. Patients with contraindications for SGM-101

     1. History of any anaphylactic shock;
     2. Patients pregnant or breastfeeding (pregnancy should be ruled out by a pregnancy test within two weeks prior to administration of the conjugate);
     3. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
     4. Previous administration of SGM-101
  2. Patients with contraindications for Indocyanine green:

     1. Allergy for shells and/or clamps
     2. Hyperthyroidism
     3. Known allergy for ICG
  3. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of simultaneous use of ICG and SGM-101 for intraoperative imaging of colorectal liver metastases. | 1.5 years
  It is deemed feasible when it meets all of the following criteria:
  1. A positive score on practical workability measured with survey A 'practical workability during surgery'
  2. A positive score on the patient's experience measured with survey B 'patient experience'.
  3. SGM-101: at least 80% sensitivity, measured as follows:
     * For capsular lesions, that are visible in white light are counted positive if TBR ≥ 1.5 in vivo.
     * For subcapsular lesions that are not visible in white light will be counted as positive if:
     A: TBR ≥ 1.5 in vivo, OR B: TBR ≥ 1.5 ex vivo on whole specimen or on bread loafs
  4. No cross-interference of fluorescent signal of both dyes within the two different excitation and emission channels.
  Feasibility is reached when a positive result on all four items is scored.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be coded and available only to the researchers of the LUMC on this particular trial. No other people will get access to the data. Results will be published.